CLINICAL TRIAL: NCT01501851
Title: Prediction of Low Birth Weight Infants Using Ultrasound Measurement of Placental Diameter and Thickness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, osama ismail kamel ibrahim, senior resident, Ain Shams Maternity Hospital
Other Study IDs: placenta and lowbirth weight
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prediction of Low Birth Weight Infants using Ultrasound Measurement of Placental Diameter and Thickness

DETAILED DESCRIPTION:
The aim of the present study is to assess the value of using ultrasound measurement of placental diameter and thickness as a predictor of low birthweight.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton viable pregnancy.
2. Gestational age at least 36 complete weeks as calculated by LMP.
3. Non scared uterus.

Exclusion Criteria:

1. Multiple fetal pregnancy.
2. Intrauterine fetal death.
3. Known congenital fetal anomalies.
4. Presence of uterine or adnexal gross pathology.
5. Presence of any medical disorder e.g. Diabetes mellitus & hypertension.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: tertiarty care clinic
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic at Ain Shams University Maternity Hospital., Cairo, Cairo Governorate, Egypt